CLINICAL TRIAL: NCT03550443
Title: RTA 402 Phase 3 Clinical Trial (A Randomized, Double-blind, Placebo-controlled Clinical Trial in Patients With Diabetic Kidney Disease)
Brief Title: A Phase 3 Study of Bardoxolone Methyl in Patients With Diabetic Kidney Disease; AYAME Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on results of double-blind parts, it was determined that it would be difficult to submit a marketing authorization application for RTA 402 for diabetic kidney disease.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 402-006
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Kidney Disease
Keywords: Bardoxolone Methyl; Diabetic Kidney Disease; Diabetes Mellitus; Kidney Diseases
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — bardoxolone methyl

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded part followed by open label extension part.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RTA 402(Bardoxolone methyl) (Experimental): Patients will receive multiple oral doses of bardoxolone methyl once daily. The starting dose of bardoxolone methyl will be 5 mg. The maximum dose will be 15 mg, and the dose will be increased by 5 mg.
  Interventions: Drug: Bardoxolone methyl
- Placebo (Placebo Comparator): Patients randomized to placebo will remain on placebo throughout the study, undergoing sham titration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bardoxolone methyl — Bardoxolone methyl 5 mg capsules
  Other Names: RTA 402
  Arms: RTA 402(Bardoxolone methyl)
Drug: Placebo — Capsules containing an inert placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of multiple oral doses of RTA 402 (5, 10, or 15 mg) administered once daily in patients with diabetic kidney disease (DKD) using the time to onset of a ≥ 30% decrease in estimated glomerular filtration rate calculated from serum creatinine (eGFR) from baseline or end-stage renal disease (ESRD) as an indicator in a randomized, double-blind, placebo-controlled study; the safety of RTA 402 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DKD
* Mean eGFR ≥ 15 and < 60 mL/min/1.73 m²
* Albumin/creatinine ratio (ACR) ≤ 3500 mg/g Cr
* Treatment with an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) with no change in dosage or medication etc.

Exclusion Criteria:

* Diabetes mellitus that is neither type 1 nor type 2
* Decreased renal function mainly attributed to a non-diabetic cause
* History of renal transplantation or upcoming preemptive renal transplantation
* Confirmed mean systolic blood pressure > 160 mmHg or a confirmed mean diastolic blood pressure > 90 mmHg during the 8-week period before screening
* Hemoglobin A1c level > 10.0% during screening
* Serum albumin level ≤ 3.0 g/dL during screening
* Cardiovascular disease specified in the study protocol
* History of cardiac failure
* BNP level > 200 pg/mL during screening etc.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1323 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Time to onset of a ≥ 30% decrease in eGFR from baseline or ESRD | Through double-blind part completion, approximately 3 to 4 years

SECONDARY OUTCOMES:
Time to onset of a ≥ 40% decrease in eGFR from baseline or ESRD | Through double-blind part completion, approximately 3 to 4 years
Time to onset of a ≥ 53% decrease in eGFR from baseline or ESRD | Through double-blind part completion, approximately 3 to 4 years
Time to onset of ESRD | Through double-blind part completion, approximately 3 to 4 years
Change in eGFR from baseline at each evaluation time point | Through double-blind part completion, approximately 3 to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Japan Community Health care Organization Sendai Hospital, Sendai, Miyagi, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoshioka K, Kaneko H, Haruyama W, Tomiyama T, Takami A, Kitayama T, Yamasaki K. Multi-Omics Reveal Antioxidant Effects of Bardoxolone Methyl in the Phase 2 Study of Bardoxolone Methyl in Patients with CKD and Type 2 Diabetes Study. Kidney360. 2025 Nov 1;6(11):1880-1889. doi: 10.34067/KID.0000000853. Epub 2025 Jun 11. PMID 40498549